CLINICAL TRIAL: NCT06177106
Title: An Assessment of Acute Solar UV-induced PD-L1/PD1 Expression in Sun Damaged & Sun Protected Human Skin of Participants With and Without History of SCC
Brief Title: SUV PDL1/PD1 in Sun Damaged & Sun Protected Human Skin of Participants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00003323; P01CA027502 (NIH)
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Other Skin Changes Due to Chronic Exposure to Nonionizing Radiation
Keywords: Sun Damaged Skin; Squamous Cell Skin Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A - history of > 2 Cutaneous squamous cell carcinoma (cSCC) (Other): Participants who have a history of squamous cell skin cancer (n=23) will be exposed to acute solar simulated light (SSL). Participants must have sun damage on the forearm, based on a standardized clinical photodamage scale (Hu C, Curiel-Lewandrowski C. Archives of Dermatology, 2011; 147(1):31-36). Each subject will act as his/her own control to minimize inter-subject variability. Subjects from each cohort will be matched based on age and gender.
  Interventions: Other: Solar Simulated Light
- Cohort B - no history of cSCC (Other): Participants without a history of squamous cell skin cancer (n=23) will be exposed to acute solar simulated light (SSL). Participants must have sun damage on the forearm, based on a standardized clinical photodamage scale (Hu C, Curiel-Lewandrowski C. Archives of Dermatology, 2011; 147(1):31-36). Each subject will act as his/her own control to minimize inter-subject variability.
  Interventions: Other: Solar Simulated Light

INTERVENTIONS:
Other: Solar Simulated Light — Acute SSL will be delivered to sun damaged skin at a rate of two-times the minimal erythema dose of each individual subject. Minimal erythema dose is defined as the smallest dose of energy necessary to produce confluent erythema with four distinct borders at 22-26 hours post-exposure.

SUMMARY:
The purpose of this research study is to look at how the proteins and genes in people's skin change when they're exposed to simulated sunlight. The researchers want to see if there are differences between people who've had skin cancer and those who haven't despite having a similar type of skin and history of sun exposure. Since this study is designed to simulate sun exposure to small areas of skin, mild to moderate sunburn and tanned spots at the site of the simulated sunlight exposure is a risk. In addition to simulated sun exposure, patients will also have four 6 mm punch skin biopsies performed. Brief discomfort may be felt when the local painkiller (lidocaine) is injected prior to skin biopsies; however, it is usually minimal. Participation in the study involves 4 visits to the clinic over the course of 4 weeks. Each visit will take no longer than 90 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals 40 years of age or older. Note: When the two groups are paired, participants will be balanced within 5 years of age. Ex. From 2.5 years younger or 2.5 years older.
* Individuals with moderate or severe photodamage of the skin on the forearms and Fitzpatrick skin type II or III (21 CFR 352.72).
* Individuals with a history of two or more cSCCs within the past 5 years (maximum of 23 enrolled) or individuals with no history of cSCC (maximum of 23 enrolled)
* Females of childbearing potential will need to undergo a pregnancy test at the enrollment visit, after administration of the ICF (informed consent form) and before exposure to solar simulated light (SSL) Premenopausal female subjects must use an effective method of birth control (such as oral contraceptives, consistent use of barrier contraceptives, IUD (intrauterine device), or other proven method of birth control) during study participation. For the purposes of this study, a woman will be considered postmenopausal if any of the following criteria are met: (1) she has had prior bilateral oophorectomy; (2) she is over the age of 60 years; or (3) she is under the age of 60 years and has not had a menstrual period in 12 or more months in the absence of chemotherapy, tamoxifen, toremifene, or ovarian suppression.
* Individuals who are willing to limit sun exposure to the body during the study period and who agree to wear protective clothing when they are outdoors.
* Individuals who have the ability to understand and willingness to sign an informed consent before initiation of study procedures, after the nature of the study is explained to them and they have had the opportunity to ask any questions.

Exclusion Criteria:

* Individuals with any inflammation or irritation of the skin at the test areas, or any skin conditions felt by the study healthcare provider to contraindicate enrollment. This includes, but is not limited to, psoriasis or atopic dermatitis within the test areas. (Test area is defined as the 6 mm areas of skin that is exposed to SSL and will be biopsied.)
* Individuals with a history of untreated skin cancer or melanocytic lesions in the test areas are ineligible. History of such conditions at a body site other than the test areas is not exclusionary if in the opinion of the study healthcare provider it will not pose a risk to the subject.
* Individuals who have had invasive cancer, chemotherapy or radiation therapy within five years of study enrollment
* Individuals who are immunosuppressed by virtue of medication or disease. This includes AIDS patients, subjects taking oral steroids, and subjects on immunosuppressants/immunomodulators (cyclosporine, chemotherapeutic agents, or biologic therapy), as determined by the examining study healthcare provider
* Individuals with serious intercurrent illness including, but not limited to, ongoing or active infection, psychiatric illness, or other situations that in the opinion of the examining study physician would limit compliance or interfere with the study regimen.
* Individuals who have used photosensitizing drugs within 30 days of enrollment, or who will be using a photosensitizing drug during the time of the study, will not be eligible.
* Individuals who have used any topical medication other than emollients or sunscreen/sunblock on the test area within 30 days prior to study enrollment. If a study participant requires topical medication to the test area during the study, they will be withdrawn from the study.
* Individuals who have used retinoids, steroids, 5-fluorouracil, Levulan, Vaniqua (eflornithine), Solaraze, or Imiquimod (Aldara®) anywhere on the body within 30 days prior to study enrollment. Subjects may be reconsidered for eligibility 30 days after the last topical treatment with such medications.
* Individuals must not take mega-doses of vitamins. Mega-doses are defined as more than 5 capsules of standard multivitamins daily or more than the Tolerable Upper Intake Levels of Vitamins, as defined by the Institute of Medicine, National Academy of Sciences. Such vitamin therapy must be discontinued at least 30 days prior to study entry.
* Individuals with a history of deliberate natural or artificial sun exposure (tanning) within 30 days of study enrollment are not eligible.
* Individuals with Fitzpatrick skin type I are ineligible, as the proposed SSL dose could result in a burn of greater than mild severity.
* Individuals with Fitzpatrick skin type IV, V or VI are ineligible, as they are unlikely to exhibit a salient response in the proposed design.
* Individuals currently enrolled in or who plan to enroll in another clinical trial. There must be a 30-day period between completing a previous study and enrolling in this study.
* Individuals with a known allergy to lidocaine are not eligible.
* Females who are pregnant or nursing.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-12-26 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess PD-L1 protein expression levels in the epidermal keratinocytes of subjects with and without a history of cutaneous squamous cell skin cancer. | Changes from baseline (pre-SSL exposure) to post-SSL exposure (at 24 hour post-exposure).
  The primary objective will be the relative increase in PD-L1 protein expression levels in the epidermal keratinocytes of subjects in two risk cohorts (Cohort A (history of > 2 cSCC) and Cohort B (no history of cSCC)) after acute solar simulated light treatment compared to unexposed skin within the same subject. Proteomic evaluation will be performed by reverse phase protein microarray and confirmatory IHC (immunohistochemistry) stain.

SECONDARY OUTCOMES:
Evaluation of CD70/CD27 protein expression analysis | Changes from baseline (pre-SSL exposure) to post-SSL exposure (at 24 hour post-exposure).
  Reverse phase protein microarray will be implemented to evaluate changes in CD70/CD27 protein expression and immunohistochemistry assays will analyze changes in these signaling pathways over time.
Spatial genomic assessment through whole transcriptomic analysis | Changes from baseline (pre-SSL exposure) to post-SSL exposure (at 24 hour post-exposure).
  Nanostring DSP (Digital Spatial Profiling). Whole transcriptomic analysis will assess these markers as well as query signaling pathways which may be differentially affected by UV in each group. The research team will perform NanoString spatial whole transcriptomic analysis on SD (sun damaged) skin samples in the 20 participants from each cohort by evaluating both pre- and post- SSL exposure, resulting in 2 matched pairs per study subject. The research team will also use DermTech RNA-seq for skin sampling and gene expression analysis on a subset of sun damaged skin samples.
High dimensional data analysis | Changes from baseline (pre-SSL exposure) to post-SSL exposure (at 24 hour post-exposure).
  The objective is to integrate the proteomic and genomic data to evaluate possible synergistic relationship between them in describing the risk of cSCC based on PD-L1/PD1 and other co-expressed genes/protein expression.

CONTACTS AND LOCATIONS:
Overall Officials: Clara Curiel-Lewandrowski, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Cancer Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided